CLINICAL TRIAL: NCT06936007
Title: Hematological Manifestations in Systemic Lupus Erythematosus: A Retrospective Cross-sectional Study From a Tertiary Care Center in Nepal
Brief Title: Hematological Manifestations in Systemic Lupus Erythematosus Patients
Status: Completed | Type: Observational
Sponsor: Patan Academy of Health Sciences (Other)
Responsible Party: Principal Investigator, Krishna Adhikari, Lecturer, Patan Academy of Health Sciences
Other Study IDs: drs2412171972
Record Dates: First submitted 2025-04-07; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: hematological manifestations; Nepal; organ involvement; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Systemic Lupus Erythematosus Patients: Patients diagnosed with systemic lupus erythematosus as per 2019 European League of Associations for Rheumatology and American College of Rheumatology (2019 EULAR/ACR) criteria

SUMMARY:
The goal of this observational study is to evaluate hematological abnormalities among patients with systemic lupus erythematosus (SLE) admitted to a tertiary care center in Nepal. The main question it aims to answer is:

- What are the types and frequencies of hematological abnormalities seen in hospitalized SLE patients in Nepal?

The study retrospectively reviews medical records of SLE patients admitted between April 2018 and March 2023 to collect data on hematologic parameters, demographic profiles, clinical manifestations.

ELIGIBILITY:
Inclusion Criteria:

* All the patient diagnosed with systemic lupus erythematosus based on 2019 European League of Associations for Rheumatology and American College of Rheumatology (2019 EULAR/ACR) criteria.

Exclusion Criteria:

* Underlying hematological diseases or conditions: Patients who had hematological disease (e.g. hemophilia, leukemia, lymphoma) or conditions that could independently affect hematological parameters.
* Incomplete records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted with diagnosis of systemic lupus erythematosus in medical ward of Patan Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with hematological abnormalities | Baseline at the time of hospital admission. (Cross-sectional)
  Anemia was defined as a Hb of less than 13 g/dL in males and less than 12 g/dL in females.
  Leukopenia was defined as a WBC of less than 4000 per cubic millimeter (cu.mm). Thrombocytopenia was defined as a platelet count of less than 100,000 per cubic millimeter.
  Lymphopenia and neutropenia were defined as absolute lymphocyte count less than 1500 per cu.mm and absolute neutrophil count less than 1800 per cu.mm.

SECONDARY OUTCOMES:
Percentage of SLE patients with mucocutaneous involvement | Through study completion from 2019 January to 2023 December.
  Proportion of patients exhibiting at least one mucocutaneous manifestation (malar rash, discoid rash, alopecia, or oral ulcers) based on physician-documented diagnosis following 2019 EULAR/ACR criteria.
Percentage of SLE patients with pericarditis | Through the study completion from 2019 January to 2023 December.
  Proportion of patients exhibiting pericarditis based on physician-documented diagnosis following 2019 EULAR/ACR criteria.
Percentage of SLE patients with respiratory involvement | Through the study completion from 2019 January to 2023 December.
  Proportion of patients exhibiting respiratory involvement based on physician-documented diagnosis following 2019 EULAR/ACR criteria.
Percentage of SLE patients with gastrointestinal involvement | Through the study completion from 2019 January to 2023 December.
  Proportion of patients exhibiting gastrointestinal involvement based on physician-documented diagnosis following 2019 EULAR/ACR criteria.
Percentage of SLE patients with kidney involvement | Through the study completion from 2019 January to 2023 December.
  Proportion of patients exhibiting kidney involvement based on physician-documented diagnosis following 2019 EULAR/ACR criteria.
Percentage of SLE patients with musculoskeletal involvement | Through the study completion from 2019 January to 2023 December.
  Proportion of patients exhibiting musculoskeletal involvement based on physician-documented diagnosis following 2019 EULAR/ACR criteria.
Percentage of SLE patients with neurological involvement | Through the study completion from 2019 January to 2023 December.
  Proportion of patients exhibiting neurological involvement based on physician-documented diagnosis following 2019 EULAR/ACR criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Patan Hospital, Lalitpur, Bagmati Province, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Systemic Lupus Erythematosus. Arthritis Rheumatol. 2019 Sep;71(9):1400-1412. doi: 10.1002/art.40930. Epub 2019 Aug 6. PMID 31385462
- [Background] Beyan E, Beyan C, Turan M. Hematological presentation in systemic lupus erythematosus and its relationship with disease activity. Hematology. 2007 Jun;12(3):257-61. doi: 10.1080/10245330701214145. PMID 17558704
- [Background] Paudyal BP, Gyawalee M. Clinical profile of patients with systemic lupus erythematosus. JNMA J Nepal Med Assoc. 2012 Jul-Sep;52(187):111-7. PMID 23591169
- [Background] Talukdar D, Gogoi A, Doley D, et al. The clinical and immunological profiles of systemic lupus erythematosus patients from Assam, North-East India. Indian J Rheumatol. 2020;15(3):181. doi:10.4103/injr.injr_37_20
- [Background] Gulati S, Kumar V, Rawat P, Chawla K, Dessai R, Jain S. Study of hematological profile of systemic lupus erythematosus. Int J Res Med Sci. 2023;11(9):3332-3335. doi:10.18203/2320-6012.ijrms20232788
- [Background] Aleem A, Al Arfaj AS, khalil N, Alarfaj H. Haematological abnormalities in systemic lupus erythematosus. Acta Reumatol Port. 2014 Jul-Sep;39(3):236-41. PMID 24861278